CLINICAL TRIAL: NCT05032950
Title: COVID-19: A PHASE 1, OPEN-LABEL, 3-TREATMENT, 6-SEQUENCE, 3-PERIOD CROSSOVER STUDY TO ESTIMATE THE EFFECT OF PF-07321332/RITONAVIR AND RITONAVIR ON THE PHARMACOKINETICS OF MIDAZOLAM IN HEALTHY PARTICIPANTS.
Brief Title: Drug-Drug Interaction Study to Estimate the Effect of PF-07321332/Ritonavir and Ritonavir on Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671013; 2021-003590-62 (EudraCT Number)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2022-12

CONDITIONS: Healthy Participants
Keywords: Drug-drug interaction; Midazolam; COVID-19 (Coronavirus disease 2019); SARS-CoV (severe acute respiratory syndrome coronavirus)
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Midazolam; nirmatrelvir; Ritonavir

STUDY DESIGN:
Intervention Model Description: This is a Phase I, crossover, 3-treatment, 6-sequence study to evaluate the effect of PF-07321332/ritonavir and ritonavir on the PK of midazolam in healthy participants. Midazolam is a substrate for CYP3A4. A total of approximately 12 healthy male and/or female participants will be enrolled into the study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Active Comparator): Midazolam orally
  Interventions: Drug: Midazolam
- Treatment B (Experimental): PF-07321332/ritonavir orally + Midazolam orally
  Interventions: Drug: PF-07321332/ritonavir + Midazolam
- Treatment C (Active Comparator): Ritonavir orally + Midazolam orally
  Interventions: Drug: Ritonavir + Midazolam

INTERVENTIONS:
Drug: Midazolam — Midazolam administered as a single dose on Day 1
  Arms: Treatment A
Drug: PF-07321332/ritonavir + Midazolam — PF-07321332/ritonavir:
  Administered orally every 12 hours for a total of 9 doses on Days 1-5
  Midazolam:
  Administered orally as a single dose on Day 5
  Arms: Treatment B
Drug: Ritonavir + Midazolam — Ritonavir:
  Administered orally every 12 hours for a total of 9 doses on Day1-5.
  Midazolam:
  Administered orally as a single dose on Day 5
  Arms: Treatment C

SUMMARY:
The purpose of this study is to estimate the effect PF-07321332/Ritonavir and Ritonavir on Midazolam (a cytochrome P450 [CYP]3A4 substrate) in Healthy Adult Participants.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants of childbearing potential must have a negative (urine or serum) pregnancy test.
2. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

   -

Exclusion Criteria:

1. Positive test result for SARS-CoV-2 infection at the time of Screening or Day -1.
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
3. Clinically relevant abnormalities requiring treatment (eg, acute myocardial infarction, unstable ischemic conditions, evidence of ventricular dysfunction, serious tachy or brady arrhythmias) or indicating serious underlying heart disease (eg, prolonged PR interval, cardiomyopathy, heart failure greater than New York Heart Association (NYHA) 1, underlying structural heart disease, Wolff Parkinson-White syndrome).
4. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
5. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or hepatitis C virus (HCVAb). Hepatitis B vaccination is allowed.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, Contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Cox DS, Rehman M, Khan T, Ginman K, Salageanu J, LaBadie RR, Wan K, Damle B. Effects of nirmatrelvir/ritonavir on midazolam and dabigatran pharmacokinetics in healthy participants. Br J Clin Pharmacol. 2023 Nov;89(11):3352-3363. doi: 10.1111/bcp.15835. Epub 2023 Jul 12. PMID 37354048
- [Derived] Sagawa K, Lin J, Jaini R, Di L. Physiologically-Based Pharmacokinetic Modeling of PAXLOVID with First-Order Absorption Kinetics. Pharm Res. 2023 Aug;40(8):1927-1938. doi: 10.1007/s11095-023-03538-5. Epub 2023 May 25. PMID 37231296
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671013

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 12 healthy participants were randomized to receive midazolam, PF-07321332/ritonavir + midazolam, and ritonavir + midazolam in a total of 6 sequences.
Groups:
- Treatment Sequence 1: Period 1: Treatment A: Midazolam Single dose of 2 mg midazolam was administered orally on Day 1, followed by serial PK sampling and 2-day washout (Duration: Day 1 to Day 3).
  Period 2: Treatment B: PF-07321332/Ritonavir + Midazolam PF-07321332 300 mg/ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
  Period 3: Treatment C: Ritonavir + Midazolam Ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
- Treatment Sequence 2: Period 1: Treatment C: Ritonavir + Midazolam Ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
  Period 2: Treatment A: Midazolam Single dose of 2 mg midazolam was administered orally on Day 1, followed by serial PK sampling and 2-day washout (Duration: Day 1 to Day 3).
  Period 3: Treatment B: PF-07321332/Ritonavir + Midazolam PF-07321332 300 mg/ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
- Treatment Sequence 3: Period 1: Treatment B: PF-07321332/Ritonavir + Midazolam PF-07321332 300 mg/ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
  Period 2: Treatment C: Ritonavir + Midazolam Ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
  Period 3: Treatment A: Midazolam Single dose of 2 mg midazolam was administered orally on Day 1, followed by serial PK sampling and 2-day washout (Duration: Day 1 to Day 3).
- Treatment Sequence 4: Period 1: Treatment C: Ritonavir + Midazolam Ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
  Period 2: Treatment B: PF-07321332/Ritonavir + Midazolam PF-07321332 300 mg/ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
  Period 3: Treatment A: Midazolam Single dose of 2 mg midazolam administered orally on Day 1, followed by serial PK sampling and 2-day washout (Duration: Day 1 to Day 3).
- Treatment Sequence 5: Period 1: Treatment B: PF-07321332/Ritonavir + Midazolam PF-07321332 300 mg/ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
  Period 2: Treatment A: Midazolam Single dose of 2 mg midazolam was administered orally on Day 1, followed by serial PK sampling and 2-day washout (Duration: Day 1 to Day 3).
  Period 3: Treatment C: Ritonavir + Midazolam Ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
- Treatment Sequence 6: Period 1: Treatment A: Midazolam Single dose of 2 mg midazolam was administered orally on Day 1, followed by serial PK sampling and 2-day washout (Duration: Day 1 to Day 3).
  Period 2: Treatment C: Ritonavir + Midazolam Ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
  Period 3: Treatment B: PF-07321332/Ritonavir + Midazolam PF-07321332 300 mg/ritonavir 100 mg was administered orally every 12 hours for a total of 9 doses on Days 1-5 and a single oral dose of midazolam 2 mg was administered on Day 5 followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
Period: Overall Study
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Treatment Sequence 3 | Treatment Sequence 4 | Treatment Sequence 5 | Treatment Sequence 6
Started (Assigned to Treatment) | 2 | 2 | 2 | 2 | 2 | 2
Completed (Completed) | 2 | 2 | 1 | 1 | 2 | 2
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants enrolled in this study
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 34.6 (9.26)
Age, Customized [Number; unit: Participants]
  <18 Years | 0
  18-25 Years | 2
  26-35 Years | 4
  36-45 Years | 4
  >45 Years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 9
  Black or African American | 1
  Asian | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Midazolam When Administered Alone and With PF-07321332/Ritonavir
Description: Cmax for midazolam following single dose administration with and without PF-07321332/ritonavir was observed directly from data. Natural log-transformed Cmax for Midazolam were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The ratios (PF-07321332/ritonavir + midazolam [test]/midazolam [reference] and 90% CIs) were expressed as percentages.
Time Frame: Midazolam: Day 1 Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 hours postdose; Midazolam+PF-07321332/ritonavir: Day 5 predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours postdose
Population: The PK parameter analysis population was defined as all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Midazolam 2 mg: Midazolam administered as a single dose on Day 1
- PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg: PF-07321332/ritonavir:
  Administered orally every 12 hours for a total of 9 doses on Days 1-5
  Midazolam:
  Administered orally as a single dose on Day 5
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 10
ng/mL | 9.812 (38) | 36.18 (17)
Statistical Analysis 1: Comparison: Midazolam 2 mg vs PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg; Natural log-transformed Cmax of midazolam was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences (AMD) (Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Reference/Test Ratio = 368.33, 90% CI 2-sided [318.91 to 425.41]

2. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 Extrapolated to Infinity Time (AUCinf) of Midazolam When Administered Alone and With PF-07321332/Ritonavir
Description: AUCinf for midazolam following single dose administration with and without PF-07321332/ritonavir was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis. Natural log-transformed AUCinf for Midazolam were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The ratios (PF-07321332/ritonavir + midazolam [test]/midazolam [reference] and 90% CIs) were expressed as percentages.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 10
ng*hr/mL | 26.13 (45) | 363.9 (13)
Statistical Analysis 1: Comparison: Midazolam 2 mg vs PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg; Natural log-transformed AUCinf of midazolam was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences (AMD) (Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Reference/Test Ratio = 1430.02, 90% CI 2-sided [1204.54 to 1697.71]

3. Primary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to the Time of the Last Quantifiable Concentration (Clast) (AUClast) of Midazolam When Administered Alone and With PF-07321332/Ritonavir
Description: AUClast for midazolam following single dose administration with and without PF-07321332/ritonavir was calculated by Linear/Log trapezoidal method. Natural log-transformed AUClast for Midazolam were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The ratios (PF-07321332/ritonavir + midazolam [test]/midazolam [reference] and 90% CIs) were expressed as percentages.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 10
ng*hr/mL | 25.02 (44) | 353.8 (13)
Statistical Analysis 1: Comparison: Midazolam 2 mg vs PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg; Natural log-transformed AUClast of midazolam was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences (AMD) (Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Test/Reference Ratio = 1451.78, 90% CI 2-sided [1224.42 to 1721.35]

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event was considered a TEAE if the event started during the effective duration of treatment. All events that start on or after the first dosing day and time/ start time, if collected, but before the last dose plus the lag time (28 days) were flagged as TEAEs. The algorithm did consider any events that started prior to the first dose date. Any events occurring following start of treatment or increasing in severity were counted as treatment emergent. Events that occur in a non-treatment period (for example, Washout or Follow-up) were counted as treatment emergent and attributed to the previous treatment taken.
Time Frame: Baseline up to Day 28
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Ritonavir 100 mg + Midazolam 2 mg: Participants administer Ritonavir orally every 12 hours for a total of 9 doses on Day1-5 and Midazolam orally as a single dose on Day 5, followed by serial PK sampling and a 7-day washout (Duration: Day 1 to Day 12).
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 11 | 11
Participants
  Participants with adverse events (All Causalities) | 4 | 9 | 7
  Participants with adverse events (Treatment related) | 4 | 9 | 7
  Participants with serious adverse events | 0 | 0 | 0
  Participants with severe adverse events | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: The haematological, clinical chemistry (serum) and urinalysis safety tests were assessed against the criteria specified in the sponsor reporting standards to determine if there were any clinically significant laboratory abnormalities. The assessment took into account whether each participant's baseline test result was within or outside the laboratory reference range for the particular laboratory parameter. Baseline was defined as the last planned predose measurement taken in each study period.
Time Frame: Baseline up to Day 28
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Ritonavir 100 mg + Midazolam 2 mg: Ritonavir:
  Administered orally every 12 hours for a total of 9 doses on Days 1-5
  Midazolam:
  Administered orally as a single dose on Day 5
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 11 | 11
Participants
  HEMATOLOGY - Lymphocytes/Leukocytes (%) >1.2x ULN | 0 | 0 | 1
  HEMATOLOGY - Neutrophils (10^3/mm^3) <0.8x LLN | 0 | 0 | 1
  HEMATOLOGY - Neutrophils/Leukocytes (%) <0.8x LLN | 0 | 1 | 1
  HEMATOLOGY - Eosinophils/Leukocytes (%) >1.2x ULN | 0 | 1 | 1
  HEMATOLOGY - Monocytes/Leukocytes (%) >1.2x ULN | 1 | 1 | 2
  HEMATOLOGY - Prothrombin Time (sec) >1.1x ULN | 0 | 0 | 1
  CLINICAL CHEMISTRY - Thyrotropin (uIU/mL) <0.8x LLN | 1 | 1 | 1
  CLINICAL CHEMISTRY - Fibrinogen (mg/dL) >1.25x Baseline | 1 | 1 | 0
  URINALYSIS - URINE Hemoglobin (Scalar) ≥1 | 2 | 1 | 3

6. Secondary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Baseline was the last predose recording in each study period. Only post baseline values are included in this analysis
Time Frame: Baseline up to Day 28
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 11 | 11
Participants | 0 | 1 | 0

7. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Baseline and changes from baseline in PR, QT, QRS, heart rate and QTcF were summarized by treatment and time postdose. Baseline was defined as the average of the triplicate predose recordings in each study period. ECG endpoints and changes from baseline (QTcF, PR, QRS), over all measurements taken postdose, were also summarized descriptively by treatment using categories as defined in the Criteria for Safety Values of Potential Clinical Concern appendix of the protocol and for QTc values corresponding to ICH E14 thresholds, which are: QTcF (msec): 450<value≤480; 480<value≤500; >500; QTcF (msec) increase from baseline: 30<change≤60; change>60
Time Frame: Baseline up to Day 28
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 11 | 11
Participants
  PR INTERVAL, AGGREGATE (MSEC) - Value≥300 | 0 | 0 | 0
  PR INTERVAL, AGGREGATE (MSEC) - %Change≥25/50% | 0 | 0 | 0
  QRS DURATION, AGGREGATE (MSEC) - Value≥140 | 0 | 0 | 0
  QRS DURATION, AGGREGATE (MSEC) - %Change≥50% | 0 | 0 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) - 450<Value≤480 | 0 | 0 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) - 480<Value≤500 | 0 | 0 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) - Value>500 | 0 | 0 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) - 30<Change≤60 | 0 | 0 | 0
  QTCF INTERVAL, AGGREGATE (MSEC) - Change>60 | 0 | 0 | 0

8. Secondary Outcome: Cmax of Midazolam When Administered Alone and With Ritonavir
Description: Cmax for midazolam following single dose administration with and without ritonavir was observed directly form data. Natural log-transformed Cmax for Midazolam were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The ratios (ritonavir + midazolam [test]/midazolam [reference] and 90% CIs) were expressed as percentages.
Time Frame: Midazolam: Day 1 Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 hours postdose; Midazolam/ritonavir: Day 5 predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Ritonavir 100 mg + Midazolam 2 mg: ritonavir: Administered orally every 12 hours for a total of 9 doses on Day1-5.
  Midazolam:
  Administered orally as a single dose on Day 5
Arm/Group | Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 10
ng/mL | 9.812 (38) | 38.03 (18)
Statistical Analysis 1: Comparison: Midazolam 2 mg vs Ritonavir 100 mg + Midazolam 2 mg; Natural log-transformed Cmax of midazolam was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences (AMD)(Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Test/Reference Ratio = 387.20, 90% CI 2-sided [335.25 to 447.21]

9. Secondary Outcome: AUCinf of Midazolam When Administered Alone and With Ritonavir
Description: AUCinf for midazolam following single dose administration with and without ritonavir was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis. Natural log-transformed AUCinf for Midazolam were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The ratios (ritonavir + midazolam [test]/midazolam [reference] and 90% CIs) were expressed as percentages.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 10
ng*hr/mL | 26.13 (45) | 418.6 (15)
Statistical Analysis 1: Comparison: Midazolam 2 mg vs Ritonavir 100 mg + Midazolam 2 mg; Natural log-transformed AUCinf of midazolam was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences (AMD)(Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Test/Reference Ratio = 1645.15, 90% CI 2-sided [1385.75 to 1953.11]

10. Secondary Outcome: AUClast of Midazolam When Administered Alone and With Ritonavir
Description: AUClast for midazolam following single dose administration with and without ritonavir was calculated by Linear/Log trapezoidal method. Natural log-transformed AUClast for Midazolam were analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The ratios (ritonavir + midazolam [test]/midazolam [reference] and 90% CIs) were expressed as percentages.
Time Frame: Midazolam: Day 1 Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 hours postdose; Midazolam/ritonavir: Day 5 pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36, 48 and 72 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 10
ng*hr/mL | 25.02 (44) | 408.8 (15)
Statistical Analysis 1: Comparison: Midazolam 2 mg vs Ritonavir 100 mg + Midazolam 2 mg; Natural log-transformed AUClast of midazolam was analyzed using mixed effect model with treatment, period and sequence as fixed effects and participant in sequence as random effect. Estimates of the adjusted mean differences (AMD)(Test-Reference) and 90%CIs were obtained from the model. The AMD and 90%CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90%CI for the ratios; Test type: Other; Mixed Models Analysis; Test/Reference Ratio = 1677.25, 90% CI 2-sided [1414.59 to 1988.69]

11. Secondary Outcome: Apparent Clearance (CL/F) of Midazolam When Administered Alone, With PF-07321332/Ritonavir, and With Ritonavir
Description: CL/F for midazolam following single dose administration with and without PF-07321332/ritonavir or ritonavir was calculated by Dose/AUCinf.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre/hour
Groups:
- Ritonavir 100mg+ Midazolam 2mg: Ritonavir:
  Administered orally every 12 hours for a total of 9 doses on Days 1-5
  Midazolam:
  Administered orally as a single dose on Day 5
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100mg+ Midazolam 2mg
Number analyzed (Participants) | 10 | 10 | 10
Litre/hour | 76.57 (45) | 5.500 (13) | 4.776 (15)

12. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Midazolam When Administered Alone, With PF-07321332/Ritonavir, and With Ritonavir
Description: Vz/F for midazolam following single dose administration with and without PF-07321332/ritonavir or ritonavir was calculated by Dose/(AUCinf • kel).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100mg+ Midazolam 2mg
Number analyzed (Participants) | 10 | 10 | 10
Litre | 488.6 (48) | 79.84 (28) | 76.43 (31)

13. Secondary Outcome: Time for Cmax (Tmax) of Midazolam When Administered Alone, With PF-07321332/Ritonavir, and With Ritonavir
Description: Tmax for midazolam following single dose administration with and without PF-07321332/ritonavir or ritonavir was calculated by observed directly from data as time of first occurrence.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100mg+ Midazolam 2mg
Number analyzed (Participants) | 10 | 10 | 10
Hour | 1.00 [0.500 to 1.10] | 1.00 [0.500 to 1.05] | 1.02 [0.500 to 3.17]

14. Secondary Outcome: Terminal Half-life (t1/2) of Midazolam When Administered Alone, With PF-07321332/Ritonavir, and With Ritonavir
Description: t½ for midazolam following single dose administration with and without PF-07321332/ritonavir or ritonavir was calculated by Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
Number analyzed (Participants) | 10 | 10 | 10
Hour | 4.988 (2.2058) | 10.47 (2.9096) | 11.54 (3.4741)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Arm/Group | Midazolam 2 mg | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg | Ritonavir 100 mg + Midazolam 2 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 4/10 | 9/11 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam 2 mg (N=10) | PF-07321332 300 mg/Ritonavir 100 mg + Midazolam 2 mg (N=11) | Ritonavir 100 mg + Midazolam 2 mg (N=11)
Nodal rhythm (Cardiac disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1 | 0
Vessel puncture site reaction (General disorders) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 6 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 3 | 3
Nightmare (Psychiatric disorders) | 1 | 1 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/50/NCT05032950/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT05032950/SAP_001.pdf